CLINICAL TRIAL: NCT06147232
Title: Prevention of CKD Progression in Type 1 Diabetes With Long Term Use of SGLTi Avoiding Kidney hypOxia(PLUTO)
Brief Title: Prevention of Chronic Kidney Disease(CDK) Progression in Type 1 Diabetes With Long Term Use of Sodium-Glucose-coTransporter Inhibitors Avoiding Kidney hypOxia
Acronym: PLUTO
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Steno Diabetes Center Copenhagen (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other); King's College London (Other); Glostrup University Hospital, Copenhagen (Other); Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: EUCT 2023-509450-55-00
Record Dates: First submitted 2023-11-19; First posted 2023-11-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Nephropathy; Diabetic Nephropathies; Diabetes Mellitus, Type 1; Albuminuria; Diabetic Complications Renal; Diabetic Complications Cardiovascular; Hypoxia
MeSH Terms: conditions — Kidney Diseases; Diabetic Nephropathies; Diabetes Mellitus, Type 1; Albuminuria; Hypoxia | interventions — (2S,3R,4R,5S,6R)-2-(4-chloro-3-(4-ethoxybenzyl)phenyl)-6-(methylthio)tetrahydro-2H-pyran-3,4,5-triol

STUDY DESIGN:
Intervention Model Description: randomized, double-blinded, placebo-controlled, cross-over intervention study
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- order: placebo/sotagliflozin (Experimental): first treatment period: 12 weeks placebo follow by: 6 weeks washout second treatment period: 12 weeks Sotagliflozin 200mg
  Interventions: Drug: Sotagliflozin; Drug: Placebo
- order: sotagliflozin/placebo (Experimental): first treatment period: 12 weeks Sotagliflozin 200mg follow by: 6 weeks washout second treatment period: 12 weeks placebo
  Interventions: Drug: Sotagliflozin; Drug: Placebo

INTERVENTIONS:
Drug: Sotagliflozin — Sodium-glucose-co-transporter 1 and 2 inhibitor
  Other Names: Inpefa (TM)
Drug: Placebo — Placebo tablet

SUMMARY:
Background: Sodium-glucose-cotransporter (SGLT) inhibition has been observed to reduce risk of cardiovascular events and kidney failure in persons with type 2 diabetes. People with type 1 diabetes also have increased risk of cardiovascular and kidney disease, and may benefit from SGLT-inhibition. The exact mechanism of how SGLT-inhibition benefits the kidneys are yet unknown. Change in renal hypoxia may be a factor.

Objective: The primary aim of this study is to assess the effects of 12 weeks SGLT-1 and 2 inhibition on renal oxygenation in persons with type 1 diabetes and chronic kidney disease.

Further aims are to study if renal oxygen consumption and response to SGLT-inhibition differs between people of African-Caribbean or Northern European decent.

Additionally effects on left ventricular ejection fraction, kidney function and biomarkers in blood and urine will be explored.

Method: 12 weeks treatment with oral sotagliflozin or matching placebo as intervention. Kidney oxygenation and perfusion parameters and left ventricular ejection fraction will be assessed by functional magnetic resonance imaging. Kidney function and biomarkers will be assessed according to local hospital laboratory guidelines.

Design: Randomized, double-blinded, placebo-controlled, cross over intervention study.

Study population: 69 persons with type 1 diabetes and diabetic kidney disease with albuminuria will be included, 39 at Steno Diabetes Center Copenhagen, 30 at King's College London.

Endpoints: Primary end-point: Change from 0 to 12 weeks in dynamic R2*-weighted signal after treatment with sotagliflozin compared to placebo. Secondary endpoints: Change from 0 to 12 weeks with sotagliflozin compared with placebo on renal perfusion, renal artery flow, renal oxygen consumption, renal parenchymal triglyceride fraction, renal fibrosis, left ventricular ejection fraction, urinary albumin-creatinin ratio, ketone bodies, erythropoietin, pro brain natriuretic peptide, and plasma- and urine inflammation- and fibrosis biomarkers as well as difference after 12 weeks treatment in glomerular filtration rate.

Timeframe: Inclusion of patients from february 2024. Last visit september 2025. Presentation spring 2026, publication fall 2026.

ELIGIBILITY:
Inclusion Criteria:

1. Persons ≥ 18 years of age with a diagnosis of type 1 diabetes (age at onset <40 years; permanent insulin treatment initiated within 1 year of diagnosis)
2. Albuminuria: UACR > 100 mg/g (in ≥2 out 3 morning spot urine collections prior to randomization)
3. estimated Glomerular Filtration Rate(eGFR) ≥25 and < 75 ml/min/1.73m2
4. Participants must be on stable renin-angiotensin system blocking treatment 4 weeks before start of study drug and throughout study duration.
5. Able to understand the written participant information and give informed consent

Exclusion Criteria:

1. Non-diabetic kidney disease indicated by medical history and/or laboratory findings.
2. eGFR< 25 ml/min/1.73m2, dialysis or kidney transplantation.
3. Previous diabetic ketoacidosis, except at debut.
4. Dysregulated diabetes (HbA1c > 85 mmol/mol)
5. Decreased awareness or unawareness
6. Pregnancy, lactating or with a wish of pregnancy within the next year
7. Low carbohydrate diet
8. Receiving therapy with an SGLT inhibitor within 8 weeks prior to enrolment or previous intolerance of an SGLT inhibitor.
9. New York Heart Association (NYHA) class IV Congestive Heart Failure at the time of enrolment
10. Myocardial infarction, unstable angina, stroke or transient ischemic attack within 12 weeks prior to enrolment
11. The receipt of any investigational product 90 days prior to this trial
12. Unable to participate in study procedures
13. Any clinically significant disorder, except for conditions associated with type 1 diabetes, which in the Investigators opinion could interfere with the results of the trial
14. Participation in another intervention study
15. Exclusion criteria for MRI: known claustrophobia, known chronic lung disease, surgery within past 6 weeks or having foreign bodies of metal in the body (e.g. pacemaker, metal plates, metal screws)
16. Recurrent urogenital infections.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Change in dynamic R2*-weighted signal (BOLD) as an indirect measure of renal blood oxygenation | 0 to 12 weeks in both treatment arms, last measure 30 weeks after randomization.
  difference between change from 0 to 12 weeks after treatment with sotagliflozin compared to treatment with placebo

SECONDARY OUTCOMES:
Change in renal perfusion (medullary and cortical) | From 0 to 12 weeks in each treatment arm. Last measure 30 weeks after randomization
  Measured with MRI by arterial spin labelling in mL/g/min
Change in renal artery flow | From 0 to 12 weeks in each treatment arm. Last measure 30 weeks after randomization
  Renal artery flow measured by using phase contrast (PC) MRI. It is measured in mL/min.
Change in renal oxygen consumption | From 0 to 12 weeks in each treatment arm. Last measure 30 weeks after randomization
  Renal oxygen consumption measured by MRI with T2-relaxation-under-spin-tagging.
Change in renal parenchymal triglyceride fraction | From 0 to 12 weeks in each treatment arm. Last measure 30 weeks after randomization
  Renal parenchymal triglyceride fraction is measured by MRI spectroscopy
Change in renal fibrosis | From 0 to 12 weeks in each treatment arm. Last measure 30 weeks after randomization
  Renal fibrosis is measured by MRI-derived apparent diffusion coefficient
Change in left ventricular ejection fraction | From 0 to 12 weeks in each treatment arm. Last measure 30 weeks after randomization
  Left ventricular ejection fraction is assessed by MRI
Change in albuminuria | From 0 to 12 weeks in each treatment arm. Last measure 30 weeks after randomization.
  Urinary albumin-creatinine ratio (UACR) - morning void spot urine samples collected at home by participants.
Change in levels of ketone bodies | From 0 to 12 weeks in each treatment arm. Last measure 30 weeks after randomization.
  Capillary blood ketones, possibly measured by continous ketone monitoring device
Change in plasma and urine inflammation- and fibrosis biomarkers | From 0 to 12 weeks in each treatment arm. Last measure 30 weeks after randomization.
  Measured from blood and urine samples using a commercially available panel from the company Olink. Includes 92 biomarkers.
Change in endogenous erythropoietin | From 0 to 12 weeks in each treatment arm. Last measure 30 weeks after randomization.
  Analysis on blood samples at regional hospital laboratory.
Change in pro brain natriuretic peptide | From 0 to 12 weeks in each treatment arm. Last measure 30 weeks after randomization.
  Analysis on blood samples at regional hospital laboratory.
Difference in Kidney Function after 12 weeks treatment with sotagliflozin vs placebo | From 12 to 30 weeks after randomization
  Glomerular filtration rate. At Steno Diabetes Center Copenhagen this will be measured by plasma clearance of Tc-99m diethylene-triamine-pentaacetate.

OTHER OUTCOMES:
Ethnicity | From baseline to 30 weeks.
  if African-Caribbean ethnicity is associated with any of the above secondary outcomes or baseline differences in cardio-renal disease markers/imaging measures

CONTACTS AND LOCATIONS:
Locations (2):
- Steno Diabetes Center Copenhagen, Herlev, Denmark
- Guy's and St Thomas NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No